CLINICAL TRIAL: NCT01329432
Title: Early Administration of Surfactant in Spontaneous Breathing (TAKE CARE) Versus InSurE (Intubation, Surfactant, Extubation) : A Pilot Study
Brief Title: Surfactant Administration During Spontaneous Breathing
Acronym: TAKE CARE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Gozde Kanmaz, MD, Zekai Tahir Burak Maternity Teaching Hospital, Neonatal Intensive care Unit
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-019
Record Dates: First submitted 2011-04-01; First posted 2011-04-06 (Estimated); Last update posted 2011-04-06 (Estimated); Status verified 2010-12

CONDITIONS: Pneumothorax; Pulmonary Interstitial Emphysema; Bronchopulmonary Dysplasia
Keywords: surfactant; intubation; spontaneous breathing; bronchopulmonary dysplasia
MeSH Terms: conditions — Pneumothorax; Mediastinal Emphysema; Bronchopulmonary Dysplasia | interventions — Insure Cement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- take care (Sham Comparator): In TAKE CARE procedure all premature infants who suffered from respiratory distress syndrome (RDS) received 100 mg/kg of porcine surfactant preparation via an intratracheal catheter during spontaneous breathing
  Interventions: Procedure: Take care
- InSurE (Experimental): infants treated with InSurE procedure were intubated and ventilated to receive surfactant and placed on nCPAP rapidly after surfactant administration
  Interventions: Procedure: InSurE

INTERVENTIONS:
Procedure: Take care — In TAKE CARE procedure all premature infants who suffered from respiratory distress syndrome (RDS) received 100 mg/kg of porcine surfactant preparation via an intratracheal catheter during spontaneous breathing.
  Arms: take care
Procedure: InSurE — infants treated with InSurE procedure were intubated and ventilated to receive surfactant and placed on nCPAP rapidly after surfactant administration.
  Arms: InSurE

SUMMARY:
Spontaneous breathing supported by nasal continuous positive airway pressure (nCPAP) is thought to have some advantages compared with mechanical ventilation in premature infants. In addition, early surfactant administration has been shown to be superior to delayed use. The aim of this pilot study was to describe the feasibility of TAKE CARE (early administration of surfactant in spontaneous breathing) procedure and compare its short-term and long-term results with InSurE procedure.

DETAILED DESCRIPTION:
In TAKE CARE procedure all premature infants who suffered from respiratory distress syndrome (RDS) received 100 mg/kg of porcine surfactant preparation via an intratracheal catheter during spontaneous breathing. In the control group infants treated with InSurE procedure were intubated and ventilated to receive surfactant and placed on nCPAP rapidly after surfactant administration. The procedures were compared for short-term efficacy and possible complications.

ELIGIBILITY:
Inclusion Criteria:

* All infants who presented with clinical anl laboratory signs of RDS

Exclusion Criteria:

* infants who required intubation or PPV right after birth

Ages: 23 Weeks to 35 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-01 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
nasal cPAP failure and need for mechanical ventilation within 72 hours | first 72 hours

SECONDARY OUTCOMES:
incidence of bronchopulmonary dysplasia | 8-10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Zekai tahir Burak Materntiy Teaching Hospital, Neonatal Intensive Care Unit, Ankara, Turkey (Türkiye)

REFERENCES:
- [Result] Kribs A, Hartel C, Kattner E, Vochem M, Kuster H, Moller J, Muller D, Segerer H, Wieg C, Gebauer C, Nikischin W, Wense Av, Herting E, Roth B, Gopel W. Surfactant without intubation in preterm infants with respiratory distress: first multi-center data. Klin Padiatr. 2010 Jan-Feb;222(1):13-7. doi: 10.1055/s-0029-1241867. Epub 2010 Jan 18. PMID 20084586